CLINICAL TRIAL: NCT05282914
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics Between "UI058" and "UIC202004" in Healthy Subjects
Brief Title: A Study to Compare PK, PD and Safety of UI058 and UIC202004 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI058-101
Record Dates: First submitted 2022-01-05; First posted 2022-03-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2021-02

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UI058 (Experimental)
  Interventions: Drug: administration of UI058
- UIC202004 (Active Comparator)
  Interventions: Drug: administration of UIC202004

INTERVENTIONS:
Drug: administration of UI058 — UI058 1Tab/day for 7days
  Other Names: Test
  Arms: UI058
Drug: administration of UIC202004 — UIC202004 1Tab/day for 7days
  Other Names: Reference
  Arms: UIC202004

SUMMARY:
A Study to compare pharmacokinetics, pharmacodynamics and safety of UI058 and UIC202004 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to read and understand a written informed consent, and willing to decide to participate in the study
* Healthy subjects between the ages of 19 and 55 years at screening
* Body weight more than 50.0kg(male)/45.0kg(female)
* Body Mass Index more than 18.0kg/m2 and under 30.0kg/m2

Exclusion Criteria:

* Have clinically significant disease that hepatobiliary system, kidney, respiratory system, nervous system, hemato-oncology disease, cardiovascular system
* Have a gastrointestinal disease history that can effect drug absorption or surgery
* Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of investigational product

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve within a dosing interval at steady state | Day 7, 0~24hours
  evaluation PK for Rabeprazole after multiple dose
percent change from baseline in integrated gastric acidity for 24-hour interval after 7th dose | baseline versus multiple dose during 7days
  evaluation PD for ambulatory 24hour pH monitor

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, Dr, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk national university hospital, Cheongju-si, North Chungcheong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided